CLINICAL TRIAL: NCT03525483
Title: Estimation of Glomerular Filtration Flow in Patients of Resuscitation Under Extra-bodily Assistance: Estimation Formula Versus Measured Clearance of Creatinine
Brief Title: Estimation of Glomerular Filtration Flow in Patients of Resuscitation Under Extra-bodily Assistance
Acronym: CREA-ECMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/18/0127; 2018-A00907-48 (Other: ID-RCB)
Record Dates: First submitted 2018-04-16; First posted 2018-05-15 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Extracorporeal Membrane Oxygenation Complication
Keywords: ECMO; Acute renal failure
MeSH Terms: conditions — Acute Kidney Injury | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with ECMO (Experimental): Patients with circulatory assistance by ECMO Patients are included 48 hours after ECMO VA or VV therapy and after hemodynamic stabilization defined by blood pressure stability and cardiac output for at least 12 hours without significant changes in amine flow.
  When stable they will have an Ultrasound for renal resistivity index measurement
  Interventions: Diagnostic Test: Ultrasound for renal resistivity index measurement

INTERVENTIONS:
Diagnostic Test: Ultrasound for renal resistivity index measurement — Collection of urine over 3 hours for creatinine clearance measurement, with serum creatinine in parallel with urine collection to calculate measured creatinine clearance and estimate glomerular filtration rate Evaluation of the renal vascular resistance index in Doppler ultrasound by a resuscitator trained in the technique at the time of inclusion.
  Collection of demographic, clinical and biological data for inclusion of the patient such as weight, age, sex, arterial lactatemia, arterial pH, volume status, use of diuretics, use of vasopressors, use of nephrotoxic drugs ...

SUMMARY:
The aim of the study will be to evaluate the quality of the GFR estimate of the two estimation equations (CKD-EPI and Cockcroft's formula) against the measured clearance of creatinine, which can be performed routinely in intensive care.

To determine the proportion of patients with ARC under ECMO VV or VA and determine changes in renal vascular resistance index as a function of GFR level in patients with pulsatile cardiac output.

DETAILED DESCRIPTION:
Extracorporeal assistance is recommended for patients with a potentially reversible acute risk of life that does not respond to conventional treatments. Hypoxic refractory syndromes, such as acute respiratory distress syndrome, are referred to as veno-venous ECMO (for Extracorporeal Membrane Oxygenation) (ECMO VV), whereas terminal cardiac dysfunctions require veno-arterial ECMO (VA ECMO). recovery of function (cardiotropic intoxication), or in the most severe cases, pending transplantation or long-term assistance.

This is a qualified pilot study, as it is the first one interested in evaluating the quality of the GFR estimate of the two estimation equations (CKD-EPI and Cockcroft formula) by relative to the measured clearance of creatinine, a method that can be performed routinely in intensive care, for resuscitation patients under veno-arterial or veno-venous ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* ECMO VV or VA after 48 hours of installation
* Hemodynamic stability for at least 12 hours
* Person affiliated or benefiting from a social security scheme
* Having expressed an express consent OR patient for whom a relative has given express consent

Exclusion Criteria:

* Hemodynamic instability
* Chronic renal failure patients receiving dialysis
* Need for continuous or intermittent extra-renal cleansing
* Patients under the protection of justice
* Person participating in another search including an exclusion period still in progress
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-19 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Compare the clearance of creatinine in urine with GFR | 1 hour
  Measured clearance of creatinine in urine (collected over 3 hours during haemodynamic stabilization of the patient) that will be compared to the Glomerular Filtration Rate(GFR) (estimated according to the Cockcroft and CKD-EPI formulas).

SECONDARY OUTCOMES:
Number of patients in ECMO with augmented renal clearance (ARC) | 1 hour
  In intensive care, some patients also have an often unrecognized increase in creatinine clearance. This entity named "augmented renal clearance" or ARC is defined by creatinine clearance> 150 mL / min / 1.73 m² for a woman and> 160 mL / min / 1.73 m² for a man. It is causing a decrease in the plasma concentration of certain drugs, especially antibiotics, which can lead to a therapeutic failure.
  A poor evaluation of the renal function in the intensive care unit can lead to overdoses or to underdosages of the drugs, by phenomena of hypofiltration or on the contrary of renal hyperfiltration.
Index of renal vascular resistance | 18 months
  index of renal vascular resistance obtained by Doppler ultrasound by a resuscitator trained in the technique at the time of inclusion.
Differences in the variable GFR between patients with glomerular hypofiltration | 18 months
  Differences in the variable GFR between patients with glomerular hypofiltration, normofiltration and hyperfiltrating patients with ClCr <60 mL / min / 1.73 m², and for normofiltration patients and hyperfiltrate patients it means CrCl> 150 mL / min / 1.73 m² for a woman and CrCl> 160 mL / min / 1.73 m² for a ma).

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Ruiz, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No